CLINICAL TRIAL: NCT04618406
Title: The Effect of Negative Pressure Wound Therapy on Wound Healing in Major Amputations
Brief Title: The Effect of Negative Pressure Wound Therapy on Wound Healing in Major Amputations of the Lower Limb
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHS-KI-09-2020
Record Dates: First submitted 2020-10-19; First posted 2020-11-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Negative-Pressure Wound Therapy; Amputation; Wound Heal
Keywords: Vascular disease; Diabetes; Preventive Care; Medical technology; Surgery
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PICO VAC (Experimental): PICO14 device from Smith and Nephew. It is a Single-Use Negative Pressure Wound Therapy Device that provides an effective negative pressure of -80 mmHg for 14 days. It is an easily applied all-in-one system that ensures uniform application each time it is applied. The dressing consists of 4 distinct layers that reduce the risk of skin trauma, applies equal negative pressure to the skin and manages fluid transport away from the wound through a combination of absorption and evaporation through an airlock layer. The device is approved for the treatment of open wounds, closed surgical incisions and skin grafts. Both PICO-VAC and soft dressing are applied immediately postoperatively and removed after 12 days.
  Interventions: Device: PICO VAC
- Standard care (Active Comparator): Standard care (sterile surgical silicone foam dressing and soft dressing)
  Interventions: Other: Standard care

INTERVENTIONS:
Device: PICO VAC — PICO14 device from Smith and Nephew - Off the shelf, disposable negative pressure wound therapy device. Contains sterile dressing as well as an attached small (pager-sized) suction device/canister and provides a negative pressure of -80 mmHg for 14 days.
  Other Names: PICO VAC (Smith and Nephew)
  Arms: PICO VAC
Other: Standard care — Sterile surgical silicone foam dressing and soft dressing applied immediately postoperative and removed after 12 days
  Other Names: Sterile surgical silicone foam dressing and soft dressing
  Arms: Standard care

SUMMARY:
The socioeconomic costs of problematic and delayed wound healing following lower limb amputations are enormous to the society. Lower limb amputations is one of the longest known surgical treatments, but also one of the least investigated in the field of medical science. Negative Pressure Wound Therapy (NPWT) has emerged as a great instrument to aid healing. Studies have shown that it has a positive and measurable effect on wound healing following eg. total Knee and hip replacements. The aim of this study is to evaluate the effect of a closed NPWT on incidence of postoperative wound complications, in patients undergoing lower extremity amputation.

DETAILED DESCRIPTION:
Historically lower limb amputations have been performed to treat infection or trauma, usually in the setting of war. Today however major amputations of the lower extremities (transfemoral- (TFA), knee disarticulations (KD) and transtibial amputations (TTA)) are, in developed countries, usually performed in elderly patients with untreatable vascular disease, diabetes or a combination of both. This fragile group of patients are characterized by a high degree of comorbidity, mortality and both surgical and postoperative complications; included herein problems with wound healing. The tissue is typically poorly vascularized and prone to wound break-down, infections, necrosis etc. 10-40% of patients undergoing TFA, KD or TTA have delayed wound healing and/or insufficient wound healing, resulting in problems with the aftercare, mobilization with a prosthesis and re-amputations. Recent retrospective studies show that Negative Pressure Wound Therapy (NPWT) may have beneficial effects on incisional healing following lower limb amputations. However to our knowledge it has never been reproduced in a prospective randomized controlled setting.The aim of this study is to investigate the effect of NPWT with a PICO®️ device (Smith & Nephew) on the healing of the surgical wound following TFA, KD and TTA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transfemoral, knee disarticulations and transtibial amputations by non-traumatic indication
* Uni or bilateral amputations or re-amputations

Exclusion Criteria:

* Patients undergoing traumatic amputations
* Unwilling or unable to provide informed consent
* Inability to comply with planned study procedures
* Amputations due to malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in the number of wound complications | Measured at 5 days and 2, 3 and 6 weeks
  Dehiscence (skin or fascia), seroma, lymph leak, infection (CDC surgical site infection criteria), Hematoma, Ischemia, Necrosis requiring any further local surgical treatment

SECONDARY OUTCOMES:
Number of participants requiring re-surgery | Within the first 6 weeks after surgery
  Revision surgery
Number of participants requiring re-amputation | Within the first 6 weeks after surgery
  Re-amputation

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grau Lykkeberg, MD, Principal Investigator — Hospital Sonderjylland
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belmont PJ Jr, Davey S, Orr JD, Ochoa LM, Bader JO, Schoenfeld AJ. Risk factors for 30-day postoperative complications and mortality after below-knee amputation: a study of 2,911 patients from the national surgical quality improvement program. J Am Coll Surg. 2011 Sep;213(3):370-8. doi: 10.1016/j.jamcollsurg.2011.05.019. Epub 2011 Jul 1. PMID 21723151
- [Background] Hasanadka R, McLafferty RB, Moore CJ, Hood DB, Ramsey DE, Hodgson KJ. Predictors of wound complications following major amputation for critical limb ischemia. J Vasc Surg. 2011 Nov;54(5):1374-82. doi: 10.1016/j.jvs.2011.04.048. Epub 2011 Aug 15. PMID 21840153
- [Background] Kotha V, Walter E, Stimac G, Kim P. Incisional Application of Negative Pressure for Nontraumatic Lower Extremity Amputations: A Review. Surg Technol Int. 2019 May 15;34:49-55. PMID 30472722
- [Background] Armstrong DG, Lavery LA, Boulton AJ. Negative pressure wound therapy via vacuum-assisted closure following partial foot amputation: what is the role of wound chronicity? Int Wound J. 2007 Mar;4(1):79-86. doi: 10.1111/j.1742-481X.2006.00270.x. PMID 17425550
- [Background] Sepulveda G, Espindola M, Maureira M, Sepulveda E, Ignacio Fernandez J, Oliva C, Sanhueza A, Vial M, Manterola C. [Negative-pressure wound therapy versus standard wound dressing in the treatment of diabetic foot amputation. A randomised controlled trial]. Cir Esp. 2009 Sep;86(3):171-7. doi: 10.1016/j.ciresp.2009.03.020. Epub 2009 Jul 18. Spanish. PMID 19616774
- [Background] Armstrong DG, Lavery LA; Diabetic Foot Study Consortium. Negative pressure wound therapy after partial diabetic foot amputation: a multicentre, randomised controlled trial. Lancet. 2005 Nov 12;366(9498):1704-10. doi: 10.1016/S0140-6736(05)67695-7. PMID 16291063
- [Background] Liu X, Zhang H, Cen S, Huang F. Negative pressure wound therapy versus conventional wound dressings in treatment of open fractures: A systematic review and meta-analysis. Int J Surg. 2018 May;53:72-79. doi: 10.1016/j.ijsu.2018.02.064. Epub 2018 Mar 16. PMID 29555530
- [Background] Norman G, Goh EL, Dumville JC, Shi C, Liu Z, Chiverton L, Stankiewicz M, Reid A. Negative pressure wound therapy for surgical wounds healing by primary closure. Cochrane Database Syst Rev. 2020 May 1;5(5):CD009261. doi: 10.1002/14651858.CD009261.pub5. PMID 32356396
- [Background] Karlakki S, Brem M, Giannini S, Khanduja V, Stannard J, Martin R. Negative pressure wound therapy for managementof the surgical incision in orthopaedic surgery: A review of evidence and mechanisms for an emerging indication. Bone Joint Res. 2013 Dec 18;2(12):276-84. doi: 10.1302/2046-3758.212.2000190. Print 2013. PMID 24352756
- [Background] Karlakki SL, Hamad AK, Whittall C, Graham NM, Banerjee RD, Kuiper JH. Incisional negative pressure wound therapy dressings (iNPWTd) in routine primary hip and knee arthroplasties: A randomised controlled trial. Bone Joint Res. 2016 Aug;5(8):328-37. doi: 10.1302/2046-3758.58.BJR-2016-0022.R1. PMID 27496913
- [Background] Nherera LM, Trueman P, Karlakki SL. Cost-effectiveness analysis of single-use negative pressure wound therapy dressings (sNPWT) to reduce surgical site complications (SSC) in routine primary hip and knee replacements. Wound Repair Regen. 2017 May;25(3):474-482. doi: 10.1111/wrr.12530. Epub 2017 May 3. PMID 28370637
- [Background] Fisher DF Jr, Clagett GP, Fry RE, Humble TH, Fry WJ. One-stage versus two-stage amputation for wet gangrene of the lower extremity: a randomized study. J Vasc Surg. 1988 Oct;8(4):428-33. PMID 3172378